CLINICAL TRIAL: NCT06089200
Title: Comparison of Post-operative Analgetics With Transversus Abdominis Block and Spinal Morphine for Post-Caesarean Section: A Randomised Trial Study
Brief Title: TAP Block vs Spinal Orphine for Postoperative Caesarean Section Analgetics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AN-202310.01
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversus Abdominis Plane Block (Experimental): Twenty two subjects were given postoperative block administration in the transversus abdominis area on each side with ultrasonography (USG) guidance
  Interventions: Procedure: Transversus Abdominal Plane Block
- Spinal Morphine (Active Comparator): Twenty two subjects were given additional morphine 100 µg intrathecally
  Interventions: Procedure: Spinal Morphine

INTERVENTIONS:
Procedure: Transversus Abdominal Plane Block — 20 cc of bupivacaine 0.2% was given to the transversus abdominis plane
  Arms: Transversus Abdominis Plane Block
Procedure: Spinal Morphine — 100 µg was administered intrathecally preoperatively
  Arms: Spinal Morphine

SUMMARY:
The goal of this randomized controlled trial is to compare the effect of TAP block vs spinal morphine for post caesarean section analgesics. The main questions it aims to answer are:

* Which post op analgesic method works better for patients who underwent caesarean section
* The number of additional opioid needed

ELIGIBILITY:
Inclusion Criteria:

* Indicated for caesarean section as assessed by Obstetricians
* ASA II
* Consented to be included in the study

Exclusion Criteria:

* Allergy history
* Spinal converted to general anesthesia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 44 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Length of time the patient needed the first additional opioid analgesics | 24 hours post operative
Total need for additional opioids | 24 hours post operative

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad F Maulana, MD, Principal Investigator — Faculty of Medicine Universitas Padjadjaran Bandung; Suwarman, MD, Study Director — Faculty of Medicine Universitas Padjadjaran Bandung; Osmond M Pison, MD, Study Director — Faculty of Medicine Universitas Padjadjaran Bandung; Prapanca Nugraha, MD, Study Director — Faculty of Medicine Universitas Padjadjaran Bandung
Locations (1):
- Hasan Sadikin General Hospital, Bandung, West Java, Indonesia